CLINICAL TRIAL: NCT06465940
Title: Observational Ambispective Study on HYPE Cups Associated With HIPER Liner
Status: Completed | Type: Observational
Sponsor: Societe dEtude, de Recherche et de Fabrication (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-05
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hip Arthropathy
Keywords: Total hip arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Total hip arthroplasty — Replacement of hip joint

SUMMARY:
This study intend to collect data on total hip arthroplasty performed with HYPE cups used with conventional polyethylene liner (HIPER).

Medical Device Regulation 2017/745 regulation required proper clinical data to support claims. This study is therefore intended to provide data on HYPE devices to comply with Medical Device Regulation2047/745 regulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient was an adult at surgery,
* Patient implanted with HYPE® acetabular cup and HIPER liner,
* Patient was followed-up at least once on retrospective part of the study,
* Patient's current social security affiliation is valid.

Exclusion Criteria:

* Patient refuses the use of his/her personal data,
* Patient is unable to follow surgeon's instruction or unavailable for follow-up,
* Patient with contraindication to x-rays,
* Patient not implanted with HYPE® acetabular cup and HIPER liner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient implanted in the selected investigational site with a HYPE® acetabular cup and HIPER liner between 2016 and 2018 were identified. The following selection criteria were used.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-07-07 (Actual)

PRIMARY OUTCOMES:
Functional score | per operative period to at least 2 year
  The information will be collected through questionnaires to compare preoperatively situation to last follow-up situation

SECONDARY OUTCOMES:
Patient satisfaction | per operative period to at least 2 year
  The information will be collected from patient through questionnaires to compare preoperatively situation to last follow-up situation
Safety adverse event | per operative period to at least 2 year
  Type and occurence of adverse events
Survival rate | per operative period to at least 2 year
  Kaplan-Meier survival rates of cups and liners

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de la Côte Basque, Bayonne, France